CLINICAL TRIAL: NCT07072819
Title: Crisis Diverted: Adapting Scalable Crisis Response Interventions for People Involved in a Criminal Legal System Diversion Program
Brief Title: Pilot of Training on 988 and Narcan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Henry Ford Health + Michigan State University Health Sciences (Other); Brown University (Other)
Responsible Party: Principal Investigator, Alison Athey, Behavioral Scientist, RAND
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-N0187
Record Dates: First submitted 2025-06-25; First posted 2025-07-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Suicide; Overdose Accidental; Overdose Antidote; Crisis Response Plan
Keywords: suicide; overdose; 988; naloxone
MeSH Terms: conditions — Suicide; Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crisis Ready Training (Experimental): This is an open label pilot of a new psychoeducational Intervention called the Crisis Ready Training. The intervention combines Crisis Line Facilitation and Take Home Naloxone trainings.
  Interventions: Behavioral: Crisis Ready Training

INTERVENTIONS:
Behavioral: Crisis Ready Training — Crisis Ready Training combines Crisis Line Facilitation with Take Home Naloxone training. The intervention is delivered in a group format.

SUMMARY:
This pilot study evaluates the acceptability, appropriateness, and feasibility of a new crisis response training called Crisis Ready.

DETAILED DESCRIPTION:
The study team conducted formative work to develop a new crisis response training for people involved in a law-enforcement assisted diversion program. The training, called Crisis Ready, combines an intervention that aims to promote use of 988 with a training on the use of Naloxone to reverse and overdose. The pilot aims to collect quantitative and qualitative data about the perceptions of the training among program participants and program staff.

ELIGIBILITY:
Inclusion Criteria:

* Participates in the Baltimore Crisis Response, Inc Law Enforcement Assisted Diversion Program
* Capacity to give informed consent

Exclusion Criteria:

* Unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure | Immediately following the intervention
  Participants' perspectives of the likability of the intervention. Scores range from 1 to 5, with higher scores indicating higher levels of acceptability.
Intervention Appropriateness Measure | Immediately following the intervention
  Measures the fit of the intervention for the population. Scores range from 1 to 5 with higher scores indicating higher levels of appropriateness.

SECONDARY OUTCOMES:
Knowledge and Perceptions of 988 | Immediately before and immediately after the intervention
  Measures participants' knowledge about the 988 crisis line and comfort using 988 for themselves or others. Participants report whether or not they heard of 988 before the training. Participants rate their level of comfort utilizing 988 for themselves or others on a scale from 0 to 10 with higher scores indicating higher levels of comfort.
Knowledge and Attitudes about Narcan | Immediately before and after the intervention
  Measures participants' knowledge of the overdose reversal effects of Narcan and where to get Narcan. Participants also rate their level of comfort carrying and using Narcan in a variety of circumstances; scores range from 0 to 10 with higher scores indicating higher levels of comfort.
Access to a phone | Immediately after the intervention.
  Author developed assessment of whether or not participants have access to a phone
Perceptions of the Crisis Ready Training | Immediately after the training
  Author developed qualitative assessment of perceptions of training. The measure asks, (1) "What did you like most about this training?", (2) "What else would you have liked to hear about or do in this training?", (3) "Is there anything else you would like us to know?"

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Athey, PhD, Principal Investigator — RAND; Sapna Mendon-Plasek, PhD, Principal Investigator — RAND
Locations (1):
- Baltimore Crisis Response, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative data will be stored and shared by the National Center for Health and Justice Integration for Suicide Prevention at Michigan State University.
Time Frame: Data will be shared upon completion of all study activities and maintained for a duration that complies with the policy of the National Institute on Mental Health.
Access Criteria: Data may be accessed by researchers who submit a data request proposal and are approved by the Center.
URL: https://nchats.org/